CLINICAL TRIAL: NCT03008187
Title: A Phase I/II Study of SEL24 in Patients With Acute Myeloid Leukemia
Brief Title: MEN1703 (SEL24) in Participants With Acute Myeloid Leukemia
Acronym: Diamond-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Collaborators: Medpace, Inc. (Industry); Theradex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI24-001
Record Dates: First submitted 2016-12-10; First posted 2017-01-02 (Estimated); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Relapsed/Refractory Acute Myeloid Leukemia; IDH
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (25 mg) (Experimental): Participants received MEN1703 (25 milligrams [mg]) orally once daily for 14 consecutive days in cycles of 21 days.
  Interventions: Drug: MEN1703
- Cohort 2 (50 mg) (Experimental): Participants received MEN1703 (50 mg) orally once daily for 14 consecutive days in cycles of 21 days.
  Interventions: Drug: MEN1703
- Cohort 3 (75 mg) (Experimental): Participants received MEN1703 (75 mg) orally once daily for 14 consecutive days in cycles of 21 days.
  Interventions: Drug: MEN1703
- Cohort 4 (100 mg) (Experimental): Participants received MEN1703 (100 mg) orally once daily for 14 consecutive days in cycles of 21 days.
  Interventions: Drug: MEN1703
- Cohort 5 (125 mg) (Experimental): Participants received MEN1703 (125 mg) orally once daily for 14 consecutive days in cycles of 21 days.
  Interventions: Drug: MEN1703
- Cohort 6 (150 mg) (Experimental): Participants received MEN1703 (150 mg) orally once daily for 14 consecutive days in cycles of 21 days.
  Interventions: Drug: MEN1703

INTERVENTIONS:
Drug: MEN1703 — MEN1703 given as oral capsules once daily for 14 consecutive days over a 21-day treatment cycle.
  Other Names: SEL24-B489; SEL24

SUMMARY:
The purpose of the clinical trial is to identify the maximum tolerated dose of MEN1703 and to further investigate its safety profile in participants with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Phase I/II, open-label, multi-center, dose escalation study to estimate the maximum tolerated dose of MEN1703 in participants with acute myeloid leukemia.

The clinical trial will investigate the safety profile and anti-leukemic activity of MEN1703 in participants with AML and that have no standard therapeutic options available.

The clinical trial encompasses 2 parts:

* Part 1: Ascending dose levels - the main purpose of this part of the clinical trial is to determine the highest dose of MEN1703 considered to be well tolerated.
* Part 2: Expansion cohort - the main purpose of this part of the clinical trial is to assess the safety and anti-leukemia activity of MEN1703 given at the highest tolerated dose in participant with relapsed/refractory acute myeloid leukemia, either all comers as well as harboring isocitrate dehydrogenase (IDH1/IDH2) mutations.

Participants participating to the clinical trial will take the study drug as oral capsules once daily for 14 consecutive days over a 21-day treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of AML, all comers or bearing IDH1 or IDH2 mutation (completed)
* Participant has no standard therapeutic options available and has either relapsed AML unsuitable for intensive chemotherapy, with no standard therapeutic options and/or not eligible for any approved targeted therapy or primary refractory AML unsuitable for intensive chemotherapy, with no standard therapeutic options and/or not eligible for any approved targeted therapy

Exclusion Criteria:

* Anti-cancer treatments (including cytotoxic chemotherapy, radiotherapy, hormonal therapy, biologic, immunotherapy or investigational drugs) received within 14 days or 5 half-lives for targeted therapies (whichever is shorter) before first dose of study drug (to be supplemented)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Northside Hospital, Atlanta, Georgia
  - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Italy (3):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Clinico Humanitas, Milan
  - ASST Monza - Ospedale San Gerardo, Monza
- Poland (2):
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Oddzial Hematologii z Pododdzialem Chemioterapi, Lodz
  - Institute of Haematology and Blood Transfusion, Warsaw
- Spain (3):
  - Institut Català d'Oncologia, Badalona
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinelli G, Solomon SR, Mukherjee S, Santoro A, Strickland SA, Vives S, Ravandi F, Walter RB, Cook RJ, Lech-Maranda E, Calbacho M, Wierzbowska A, Marconi G, Acuna-Cruz E, Cano-Ferri I, Bertolini F, Rzymski T, Paoli A, Merlo GM, Auriol FK, Zicari S, Galleu A, Gupta I, Montesinos P. Dual FLT3/PIM inhibitor dapolsertib in acute myeloid leukemia: results from the phase 1/2 DIAMOND-01 trial. Blood Neoplasia. 2025 Oct 24;3(1):100178. doi: 10.1016/j.bneo.2025.100178. eCollection 2026 Feb. PMID 41536779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened across 4 countries: Unites States, Italy, Spain, and Poland.
Period: Part 1: Dose Escalation
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Started | 2 | 3 | 3 | 6 | 7 | 4
Received at Least 1 Dose of Study Drug (Safety Population) | 2 | 3 | 3 | 6 | 7 | 4
Completed | 2 | 3 | 3 | 6 | 7 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Dose Expansion
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Started | 0 (Participants from Part 1 did not carry over to Part 2.) | 0 (Participants from Part 1 did not carry over to Part 2.) | 0 (Participants from Part 1 did not carry over to Part 2.) | 0 (Participants from Part 1 did not carry over to Part 2.) | 48 (Participants from Part 1 did not carry over to Part 2.) | 0 (Participants from Part 1 did not carry over to Part 2.)
Received at Least 1 Dose of Study Drug (Safety Population) | 0 | 0 | 0 | 0 | 48 | 0
Completed | 0 | 0 | 0 | 0 | 48 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of MEN1703.
Groups:
- Cohort 1 (25 mg): Participants received MEN1703 (25 mg) orally once daily for 14 consecutive days in cycles of 21 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg) | Total
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 55 | 4 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.50 (31.820) | 71.00 (5.000) | 75.33 (8.963) | 65.67 (18.726) | 65.55 (12.060) | 63.50 (7.047) | 65.58 (12.923)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 24 | 1 | 33
  Male | 1 | 1 | 1 | 3 | 31 | 3 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 2 | 3 | 3 | 6 | 53 | 4 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 1 | 0 | 4
  White | 1 | 3 | 3 | 4 | 51 | 4 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and Part 2: Number of Participants Experiencing Treatment-emergent Adverse Events
Description: An adverse event (AE) was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the investigational medicinal product. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse events module.
Time Frame: Up to 21 months
Population: Safety population: all participants that received at least 1 dose of MEN1703.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 55 | 4
Participants | 2 | 3 | 3 | 6 | 54 | 4

2. Primary Outcome: Part 1: Number of Participants Experiencing Dose-limiting Toxicity (DLT)
Description: AEs were graded according to the National Cancer Institute common terminology criteria for adverse events, version 4.03. The following AEs were considered as DLT unless they were clearly and incontrovertibly attributable to the underlying disease or to an extraneous cause: Grade 5 toxicity; Grade 4 neutropenia lasting ≥42 days from the start of the therapy cycle in absence of evidence of active acute myeloid leukemia (AML) (<5% blasts); Grade 3 or 4 non-hematologic toxicity (with protocol-define exceptions). Only clinically significant abnormalities in laboratory findings, physical examination, vital signs, weight, or electrocardiogram were considered for DLT assessment.
Time Frame: Day 1 through Day 21 (first treatment cycle)
Population: Safety Population: all participants that received at least one dose of MEN1703. Here, 'Overall Number of Participants Analyzed' signifies those participants from Part 1 who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 7 | 4
Participants | 1 | 0 | 0 | 0 | 1 | 3

3. Secondary Outcome: Part 1 and Part 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a complete remission (CR), complete remission with incomplete hematologic recovery (CRi), complete remission with partial hematologic recovery (CRh), or morphologic leukemia-free state (MLFS) response to therapy.
Time Frame: Up to 32 months
Population: Efficacy Population: all participants in each cohort that have completed 1 cycle of treatment (considering both the treatment and the washout period) and have taken at least 75% of the study drug during the first cycle. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this Outcome Measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 37 | 2
percentage of participants |  | 0 | 50.0 | 0 | 13.5 | 0

4. Secondary Outcome: Part 1 and Part 2: Partial Remission (PR) Rate
Description: PR rate was defined as the percentage of participants who had a partial remission response to therapy.
Time Frame: Up to 32 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 37 | 2
percentage of participants |  | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Part 1 and Part 2: Duration of Response (DoR)
Description: DoR was defined as the time from the date of first CR, CRi, CRh, CR without minimal residual disease (CRMRD-), MLFS or PR until the date of documented relapse of any type, progressive disease or death due to disease progression for participants who achieve CR, CRi, CRh, CRMRD-, MLFS or PR. Results are reported in days.
Time Frame: Up to 32 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 37 | 2
days |  | NA [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). | 79.0 [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). Only 1 participant had a response. As a consequence, the standard deviation was 0 and the confidence interval limits were not estimable. | NA [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). | 63.0 [44.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events). | NA [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events).

6. Secondary Outcome: Part 1 and Part 2: Relapse Free Survival (RFS)
Description: RFS was defined as the time from the date of first CR, CRi, CRh, or CRMRD- until the date of documented relapse or death from any cause. Results are reported in days.
Time Frame: Up to 32 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 37 | 2
days |  | NA [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). | 81.0 [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). Only 1 participant had a response. As a consequence, the standard deviation was 0 and the confidence interval limits were not estimable. | NA [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). | 64.0 [44.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events). | NA [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events).

7. Secondary Outcome: Part 1 and Part 2: Overall Survival (OS)
Description: OS was defined as the number of days between the first study drug administration and death from any cause. Results are reported in days.
Time Frame: Up to 32 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 37 | 2
days |  | 43.0 [NA to NA] — NA = Values were non-estimable because the standard error was non-estimable due to an insufficient number of participants with events. | 138.5 [63.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events). | NA [108.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events). | 144.0 [72.0 to 287.0] | 42.5 [34.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events).

8. Secondary Outcome: Part 1 and Part 2: Event Free Survival (EFS)
Description: EFS was defined as the time from the date of first study drug intake until the date of documented relapse, treatment failure, or death from any cause. Results are reported in days.
Time Frame: Up to 32 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 37 | 2
days |  | 15.0 [NA to NA] — NA = Values were non-estimable because the standard error was non-estimable due to an insufficient number of participants with events. | 14.0 [NA to NA] — NA = Values were non-estimable (insufficient number of participants with events). The 2 participants with a measurable outcome reported the same result. As a consequence, standard deviation was 0 and the confidence interval limits were not estimable. | 14.0 [14.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events). | 43.0 [42.0 to 49.0] | 15.0 [14.0 to NA] — NA = Values were non-estimable (insufficient number of participants with events).

9. Secondary Outcome: Part 1 and Part 2: Transfusion Conversion Rate
Description: Transfusion conversion rate was defined as the percentage of participants who were transfusion dependent at baseline but became transfusion independent post-baseline. Participants were classified as baseline transfusion independent if there were no red blood cells (RBC) or platelet transfusions at baseline; otherwise, the participant was considered as baseline transfusion dependent. Participants were classified post-baseline transfusion independent in the event of 56 consecutive days without any RBC or platelet transfusion post-baseline; otherwise, the participant was considered post-baseline transfusion dependent.
Time Frame: Up to 21 months
Population: Efficacy Population: all participants in each cohort that have completed 1 cycle of treatment (considering both the treatment and the washout period) and have taken at least 75% of the study drug during the first cycle. Here, 'Overall Number of Participants Analyzed' signifies those participants who were transfusion dependent at baseline and had transfusion status reported post baseline. Data was collected only for Cohort 5 for this end point as pre-specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 5 (125 mg)
Number analyzed (Participants) | 4
percentage of participants | 25

10. Secondary Outcome: Part 1 and Part 2: Transfusion Maintenance Rate
Description: Transfusion maintenance rate was defined as the percentage of participants who were transfusion independent at baseline and still maintained to be transfusion independent post-baseline. Participants were classified as baseline transfusion independent if there were no RBC or platelet transfusions at baseline; otherwise, the participant was considered as baseline transfusion dependent. Participants were classified post-baseline transfusion independent in the event of 56 consecutive days without any RBC or platelet transfusion post-baseline; otherwise, the participant was considered post-baseline transfusion dependent.
Time Frame: Up to 21 months
Population: Efficacy Population: all participants in each cohort that have completed 1 cycle of treatment (considering both the treatment and the washout period) and have taken at least 75% of the study drug during the first cycle. Here, 'Overall Number of Participants Analyzed' signifies those participants who were transfusion independent at baseline and had transfusion status reported post baseline. Data was collected only for Cohort 5 for this end point as pre-specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 5 (125 mg)
Number analyzed (Participants) | 2
percentage of participants | 100

11. Secondary Outcome: Part 1 and Part 2: Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) Rate
Description: Allogeneic HSCT rate was defined as the percentage of participants undergoing allogeneic stem cell transplant during the study period of each participant.
Time Frame: Up to 21 months
Population: Efficacy Population: all participants in each cohort that have completed 1 cycle of treatment (considering both the treatment and the washout period) and have taken at least 75% of the study drug during the first cycle. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. Data was collected only for Cohort 5 for this end point as pre-specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 5 (125 mg)
Number analyzed (Participants) | 37
percentage of participants | 2.7

12. Secondary Outcome: Part 1 and Part 2: Percentage of Participants With ≥ 50% Bone Marrow Blast Reduction
Description: Bone marrow aspirates/biopsies were taken at designated timepoints for evaluation of leukemic blast proportion in the bone marrow. A reduction in bone marrow blast proportion indicates increased anti-leukemic activity of the study drug.
Time Frame: Up to 20 months
Population: Efficacy Population: all participants in each cohort that have completed 1 cycle of treatment (considering both the treatment and the washout period) and have taken at least 75% of the study drug during the first cycle. Here, 'Overall Number of Participants Analyzed' signifies those participants who had an available baseline bone marrow assessment and at least 1 post-baseline bone marrow assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 0 | 1 | 2 | 4 | 24 | 2
percentage of participants |  | 0 | 50.0 | 0 | 33.3 | 0

13. Secondary Outcome: Part 1 and Part 2: Maximum Observed Concentration (Cmax) for MEN1703
Description: Nominal blood samples were taken at designated timepoints for evaluation of concentration levels of MEN1703 in plasma. Results are reported as nanograms/milliliter (ng/mL). Standard error not reported, arithmetic coefficient of variation (CV%) reported instead.
Time Frame: Day 1 and Day 14 of Cycle 1 (pre-dose, up to 120 hours post dose) (21 days/cycle)
Population: Pharmacokinetics (PK) Population: all participants who received any dose of MEN1703 and had at least 1 measurable drug concentration. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 55 | 4
ng/mL
  Cycle 1 Day 1 | 8.77 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 29.3 | 33.58 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 33.5 | 60.55 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 88.3 | 73.25 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 50.4 | 152.94 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 54 | 249.00 (NA) — Standard error not reported, arithmetic CV% reported instead.CV% = 26.8
  Cycle 1 Day 14: number analyzed (Participants) | 0 | 3 | 3 | 6 | 42 | 3
  Cycle 1 Day 14 |  | 74.32 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 64.1 | 167.08 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 60.9 | 294.25 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 53.5 | 507.18 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 44 | 759.36 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 97.8

14. Secondary Outcome: Part 1 and Part 2: Area Under the Concentration Versus Time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) for MEN1703
Description: Nominal blood samples were taken at designated timepoints for evaluation of concentration levels of MEN1703 in plasma. AUClast was calculated by the linear trapezoidal rule. Results are reported in hour times nanograms/milliliter (h*ng/mL). Standard error not reported, arithmetic CV% reported instead.
Time Frame: Day 1 of Cycle 1 (pre-dose, up to 24 hours post dose) (21 days/cycle)
Population: Pharmacokinetics (PK) Population: all participants who received any dose of MEN1703 and had at least 1 measurable drug concentration. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Error); unit: h*ng/mL
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 55 | 4
h*ng/mL | 152.17 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 43 | 490.37 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 24.3 | 729.48 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 116.3 | 1016.62 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 69.5 | 1936.61 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 64.2 | 2608.31 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 47

15. Secondary Outcome: Part 1 and Part 2: Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours (AUC0-24) for MEN1703
Description: Nominal blood samples were taken at designated timepoints for evaluation of concentration levels of MEN1703 in plasma. AUC0-24 was calculated by the linear trapezoidal rule. Results are reported in h*ng/mL. Standard error not reported, arithmetic CV% reported instead.
Time Frame: Day 14 of Cycle 1 (pre-dose, up to 120 hours post dose) (21 days/cycle)
Population: Pharmacokinetics (PK) Population: all participants who received any dose of MEN1703 and had at least 1 measurable drug concentration. Here, 'Overall Number of Participants Analyzed' signifies those participants in Cohorts 2-6 who were evaluable for this outcome measure at the specified time point. Data was not collected for Cohort 1 for this outcome measure.
Measure: Mean (Standard Error); unit: h*ng/mL
Arm/Group | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
Number analyzed (Participants) | 3 | 3 | 6 | 38 | 3
h*ng/mL | 1330.03 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 78.4 | 2885.33 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 66.7 | 5574.10 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 52.6 | 9224.62 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 50.6 | 15769.60 (NA) — Standard error not reported, arithmetic CV% reported instead. CV% = 106.3

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to 21 months. All-cause mortality, survival (RFS, EFS, OS), ORR, PR rate, and DOR were assessed up to 32 months.
Description: All reported safety data based upon the Safety Population: all participants that received at least 1 dose of MEN1703.
Arm/Group | Cohort 1 (25 mg) | Cohort 2 (50 mg) | Cohort 3 (75 mg) | Cohort 4 (100 mg) | Cohort 5 (125 mg) | Cohort 6 (150 mg)
All-Cause Mortality (participants affected / at risk) | 2/2 | 3/3 | 3/3 | 1/6 | 35/55 | 4/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 3/3 | 6/6 | 35/55 | 4/4
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 3/3 | 6/6 | 52/55 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (25 mg) (N=2) | Cohort 2 (50 mg) (N=3) | Cohort 3 (75 mg) (N=3) | Cohort 4 (100 mg) (N=6) | Cohort 5 (125 mg) (N=55) | Cohort 6 (150 mg) (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 8 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyphaema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 17 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 5 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1 (25 mg) (N=2) | Cohort 2 (50 mg) (N=3) | Cohort 3 (75 mg) (N=3) | Cohort 4 (100 mg) (N=6) | Cohort 5 (125 mg) (N=55) | Cohort 6 (150 mg) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 3 | 17 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 7 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 6 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 13 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adrenal mass (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 9 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 7 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 26 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 4 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 13 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 19 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 1 | 3 | 7 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2 | 6 | 2
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 5 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Superinfection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0/1 | 0/2 | 1/2 | 0/3 | 0/24 | 0/1 — This adverse event affected only female participants.
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1 | 3 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 9 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 13 | 2
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 7 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1 | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 4 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 3 | 4 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 3 | 4 | 0
Prothrombin level increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 2 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 3 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 6 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 8 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 7 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 6 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 3 | 3 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal cord oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flat affect (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 4 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Vulval ulceration (Reproductive system and breast disorders) | 0/1 | 0/2 | 0/2 | 0/3 | 1/24 | 0/1 — This adverse event affected only female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study cannot be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A. has reviewed/commented and agreed to any publication.

DOCUMENTS (2):
  • Study Protocol (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03008187/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT03008187/SAP_001.pdf